CLINICAL TRIAL: NCT02170298
Title: Effects of Lisdexamfetamine on Cognitive Control and Reward Response in Adolescents and Young Adults With ADHD: Neural and Clinical Outcomes
Brief Title: Lisdexamfetamine's Effect In ADHD in the Brain and Cognition
Acronym: LEIA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of California, Davis (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 402395
Record Dates: First submitted 2014-06-11; First posted 2014-06-23 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; Vyvanse; Lisdexamfetamine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants may be randomized into the placebo comparator arm. Participants in this group will be given a sugar pill titrated up to 70 mg daily over the course of 9 weeks.
  Drug: Placebo
  Interventions: Drug: Lisdexamfetamine
- Lisdexamfetamine (Experimental): Participants may be randomized into the experimental arm. Participants in this arm will be given lisdexamfetamine titrated up to 70 mg daily over the course of 9 weeks.
  Drug: Lisdexamfetamine
  Interventions: Drug: Lisdexamfetamine

INTERVENTIONS:
Drug: Lisdexamfetamine — Participants will be given either the study drug or placebo in tablet form. All participants will start with a 20 mg dose and will be titrated up to a 70 mg daily dose over 9 weeks. Participants between 12-18 years of age will be titrated in 10 mg increments and participants between 18-25 years of age in 10-20 mg increments.
  Other Names: Vyvanse

SUMMARY:
The purpose of this study is to identify the effects of lisdexamfetamine (LDX) on the neural and behavioral subcomponents of self-control, that is cognitive control and reward functioning, in adolescents and young adults with attention-deficit/hyperactivity disorder.

The investigators hypothesize that LDX is associated with 1a) decreased task-independent locus coeruleus (LC) activity; 1b) increased task-related activity in LC and the cognitive control network; 2) increased LC connectivity with the cognitive control network and 3) improved task performance and self-control. The investigators will test their hypotheses on fMRI data with linear contrasts of voxel-wise maps of parameter estimates (in both univariate and connectivity analyses).

The investigators will also assess change in brain activity with the LDX in the LC and ventral tegmental areas (VTA) as we hypothesize that they are altered in ADHD and related to cognitive control and self-control dysfunction in ADHD.

The investigators will use a repeated-measures, between-subject design to compare the effects of oral once daily LDX in a double-blind placebo-controlled randomized trial (RCT) on neural (fMRI) and behavioral correlates of cognitive control via a working memory and a reward - delay discounting task in adolescents and young adults.

A new condition has been added which will use a within-subject comparison, cross-over design between a single dose of LDX versus a single dose of placebo.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male or female adolescent or young adult, between the ages of 12 and 30 (inclusive) at the time of the initial signing of the informed consent/assent
2. The subject meets DSM Fifth edition (DSM-5) diagnostic criteria for Attention Deficit-Hyperactivity Disorder, Combined-Type. Diagnostic Interviews and Rating Scales will be used to inform about DSM criteria. Participants with 4 or 5 hyperactive/impulsive symptoms may be included at the investigator's discretion.
3. This includes a history of childhood symptoms of ADHD for the adult subjects
4. The subject, a caregiver, and the investigator must all agree that the present ADHD symptoms cause impairment in the subject's normal routines, which include academic achievement, occupational functioning, social activities, and/or relationships
5. Females of childbearing potential (defined by menarche and not having undergone surgical sterilization/hysterectomy) must have a negative pregnancy test, must be practicing acceptable methods of contraception (or can confirm abstinence at each scheduled visit), and must not be pregnant or lactating at any point while they are participating in the study.
6. Written informed consent must be obtained from a legally acceptable representative (e.g. guardian or caregiver for minors), in accordance with requirements of the Institutional Review Board (IRB), prior to the initiation of any protocol-required procedures. In addition, the subject, as required by the IRB, must provide informed assent at screening and as such must be able to understand that he or she can withdraw from the time at any time.
7. The subject and the designated guardian(s) or caregiver(s)[If minors] are able to comprehend and satisfactorily comply with the protocol requirements, as evaluated by the investigator

Exclusion Criteria:

* Clinical contraindications

  1. History of schizophrenia, bipolar disorder, autism spectrum disorder, specific or focal neurological disorder
  2. Current academic learning disorder(s)
  3. Abnormal cardiac functioning with be excluded
  4. The subject experiences Adverse Events during the trial that would, in the investigator's judgment, preclude further exposure to LDX
  5. The subject had protocol violations during the trial considered major in the judgment of the investigator (significant noncompliance, use of prohibited concomitant medications, concern with use of drugs of abuse, etc.), which would deem them poor candidates for this trial
  6. Sexually active males who will not commit to utilizing an approved birth control methods or who will not remain abstinent during the trial and for 90 days following the last dose of study drug. Sexually active females of childbearing potential who will not commit to utilizing 1 of the approved birth control methods or who will not remain abstinent during the trial and for 30 days following the last dose of study drug. Abstinence will be permitted if it is confirmed and documented at every trial visit. If employing birth control, 1 of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pill, birth control depot injections, implant, condom or sponge with spermicide.
  7. Subjects with an inability to swallow tablets or tolerate oral medication
  8. It is in the investigator's opinion that it is not in the subject's best interest to continue
  9. Contraindication for MRI scanning (e.g., metal implants, pacemakers, metal foreign bodies, pregnancy)
* Beast-feeding (if applicable)

  1. Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving trial drug
* Excluded medications

  1. Agents that lower blood levels of amphetamines: urinary acidifying agents (e.g. ammonium chloride, sodium acid phosphate, etc.); Methenamine Therapy.
  2. Agents that increase blood levels of amphetamines: urinary alkalinizing agents (e.g. Acetazolamide, some Thiazides).
  3. Dextroamphetamine is known to inhibit monoamine oxidase, as well as a metabolite of furazolidone. Concurrent administration of monoamine oxidase (MAOI) inhibitors is contraindicated because MAOIs potentially can result in hypertensive crisis. Vyvanse should not be given for at least 14 days after discontinuation of an MAO inhibitor.
  4. Agents whose effects may be reduced by amphetamines: Adrenergic blockers, Antihistamines, Antihypertensives, Veratrum Alkaloids, Ethosuximide.
  5. Agents whose effects may be potentiated by amphetamines: Tricyclic antidepressants, meperidine, Norepinephrine, Phenobarbital, Phenytoin.
  6. Agents that may reduce the effects of amphetamines: Antipsychotics, Lithium Carbonate
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation

  1. Previous negative history with LDX
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements

  1. A positive drug screen for cocaine or other drugs of abuse (excluding caffeine, nicotine or prescribed psychostimulants for ADD/ADHD)
  2. History of substance dependence or abuse disorder currently or within past 5 years.
* Recent serious illness requiring systemic treatment and/or hospitalization prior to entry.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie B Schweitzer, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants may be randomized into the placebo comparator arm. Participants in this group will be given a sugar pill titrated up to 70 mg daily over the course of 9 weeks.
  Drug: Placebo
  Lisdexamfetamine: Participants will be given either the study drug or placebo in tablet form. All participants will start with a 20 mg dose and will be titrated up to a 70 mg daily dose over 9 weeks. Participants between 12-18 years of age will be titrated in 10 mg increments and participants between 18-25 years of age in 10-20 mg increments.
- Lisdexamfetamine: Participants may be randomized into the experimental arm. Participants in this arm will be given lisdexamfetamine titrated up to 70 mg daily over the course of 9 weeks.
  Drug: Lisdexamfetamine
  Lisdexamfetamine: Participants will be given either the study drug or placebo in tablet form. All participants will start with a 20 mg dose and will be titrated up to a 70 mg daily dose over 9 weeks. Participants between 12-18 years of age will be titrated in 10 mg increments and participants between 18-25 years of age in 10-20 mg increments.
Period: Overall Study
Arm/Group | Placebo | Lisdexamfetamine
Started | 1 | 5
Completed | 0 | 4
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — unblinded, rerandomized to intervention | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lisdexamfetamine | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Working Memory
Description: Working memory performance, as measured by the percent of items correct on the Span Working Memory Task.
Time Frame: Baseline, 9 weeks
Population: Data were not analyzed due to early study termination. Unable to recruit a sufficient number of subjects. Data on this measure is highly variable and low subject numbers will not produce reliable or valid data.
Arm/Group | Placebo | Lisdexamfetamine
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Delay Discounting
Description: Level of self-control, as demonstrated on the Delay Discounting Task.
Time Frame: Baseline, 9 weeks
Population: as for outcome 1
Arm/Group | Placebo | Lisdexamfetamine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Placebo | Lisdexamfetamine
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4

LIMITATIONS AND CAVEATS:
Data were not analyzed due to early study termination. Unable to recruit a sufficient number of subjects. Data on this measure is highly variable and low subject numbers will not produce reliable or valid data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes